CLINICAL TRIAL: NCT03138083
Title: A Modular, Multi-arm, Multi-part, First Time in Patient Study to Evaluate the Safety and Tolerability of OMO-1, Alone and in Combination With Anti-cancer Treatments, in Patients With Locally Advanced, Unresectable or Metastatic Solid Malignancies
Brief Title: OMO-1 in Solid Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: strategic reasons (not due to lack of efficacy or safety issues)
Sponsor: Octimet Oncology N.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OMO1.01.02
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Neoplasms
Keywords: Mesenchymal-epithelial transition factor (MET) inhibitor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A modular, multi-arm, multi-part, first time in patient study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Module 1 Monotherapy Multiple Ascending Dose (Experimental): Multiple ascending dose cohorts dosing OMO-1 (bid) monotherapy in all comer patients up to a maximally tolerated or maximally feasible dose
  Interventions: Drug: OMO-1
- Module 1 Monotherapy Paired Biopsy (Experimental): Paired biopsy cohort(s) dosing OMO-1 (bid) monotherapy in patients selected for MET dependent tumours at minimally biologically active doses and above
  Interventions: Drug: OMO-1
- Module 1 Monotherapy Expansion Cohort(s) (Experimental): Expansion cohort(s) dosing OMO-1 (bid) monotherapy in patients selected for MET dependent tumours at recommended phase 2 dose (RP2D)
  Interventions: Drug: OMO-1
- Module 2 Combination with EGFR-TKI Multiple Ascending Dose (Experimental): Multiple ascending dose cohorts dosing OMO-1 (bid) in combination with EGFR-TKI in MET amplified patients up to a maximally tolerated or maximally feasible dose
  Interventions: Drug: OMO-1
- Module 2 Combination with EGFR-TKI Paired Biopsy (Experimental): Paired biopsy cohort(s) dosing OMO-1 (bid) in combination with EGFR-TKI in MET amplified patients at minimally biologically active doses and above
  Interventions: Drug: OMO-1
- Module 2 Combination with EGFR-TKI Expansion Cohort (Experimental): Expansion cohort dosing OMO-1 (bid) monotherapy in combination with EGFR-TKI in MET amplified patients at recommended phase 2 (combination) dose (RP2D)
  Interventions: Drug: OMO-1

INTERVENTIONS:
Drug: OMO-1 — OMO-1 is a small molecule inhibitor of the enzymatic activity of the MET receptor tyrosine kinase
  Other Names: JNJ-38877618

SUMMARY:
This is a modular, first time in patient, open-label, multicentre study of OMO-1, administered orally, alone and in combination with anti-cancer treatments, in patients with locally advanced, unresectable or metastatic solid malignancies.

DETAILED DESCRIPTION:
The study will consist of a number of study modules. The initial Module 1 will evaluate OMO-1 as monotherapy to provide dose(s) and schedule(s) for further Modules of combination therapy.

Module 2 will evaluate OMO-1 in combination with small molecule EGFR-TKIs.

Study modules will consist of a Part A (dose finding) and an optional Part B (cohort expansion). The option to start Part B and add further modules will be the decision of the safety review committee, based on emerging preclinical anti-tumour data and, safety and tolerability information from the study as a whole.

For all modules, Part A cohorts may be expanded by up to 12 additional patients at doses (at or above the MBAD) that have been confirmed to be tolerated. These patients will have mandatory paired biopsies to assess the tumour for relevant PDc biomarkers, and to explore further the tolerability, safety and PK activity at these doses.

In all combination modules, the dose of each combination agent investigated will not exceed their current recommended dose. The starting dose of OMO-1 in combination modules will not exceed the one currently tolerated in Module 1 (monotherapy). For cohorts in which OMO-1 is dosed in combination with cytotoxic chemotherapy, dosing will not continue once the cycles of chemotherapy have been completed.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years
* Provision of signed and dated, written informed consent.
* Histological or cytological confirmation of locally advanced, unresectable or metastatic solid malignancy.
* Performance status: Eastern Co-operative Oncology Group (ECOG) ≤1 and life expectancy ≥3 months.
* Ability to swallow and retain oral medication.
* Adequate organ functions.
* Females of child-bearing potential:

  * Must use a highly effective method contraceptive measures during the study and for 1 month after the last dose of OMO 1.
  * Must not be breast feeding.
  * Must have a negative pregnancy test prior to start of dosing.
* Sexually active male patients must be willing to use barrier contraception

Exclusion Criteria:

* Patients receiving other cancer therapy, or other investigational product apart from the combination agent(s) described in the relevant combination modules.
* Patients who have received radiotherapy for the primary tumour within 1 week from the screening visit.
* Patients receiving medications predominantly metabolized by CYP2B6.
* Patients receiving cannabinoid substances.
* Patients receiving St John's Wort.
* Patients receiving medications that are known to have potent aldehyde oxidase (AO) inhibitory activity.
* Patients with prior splenectomy.
* Patients testing positive for human immunodeficiency virus (HIV) infection, hepatitis B based on findings of persistent hepatitis B virus surface antigen (HBsAg) or other serology test, hepatitis C virus (HCV) or Epstein-Barr Virus (EBV) infection.
* Patients with current, or a history of uveitis.
* Patients with any known uncontrolled inter-current illness including ongoing or active infections, symptomatic congestive heart failure, conditions that could adversely be affected by hypertension or tachycardia, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a history or clinical evidence of neoplastic central nervous system (CNS) involvement if not stable for 9 weeks prior to the first dose of study treatment.
* Patients with major and/or planned surgery within 12 weeks of the first dose of study treatment.
* Patients with any known severe allergies (e.g., anaphylaxis) to any active or inactive ingredients in OMO-1.
* Patients with nephrolithiasis.
* Patients with current, or a history of any seizure or seizure disorder. This includes receiving, or having received, seizure threshold-raising medication for the treatment of epilepsy.

In addition to the main core eligibility criteria, Module specific eligibility criteria include:

Module 1:

Patient recruited into the paired biopsy cohorts of Part A must have:

* at least 1 lesion suitable for biopsy.
* tumours that are MET gene amplified and/or mutated.
* had no prior therapy with a selective MET inhibitor.

Patients recruited into Part B cohorts must have:

* tumours that are MET gene amplified and/or mutated.
* at least one lesion, not previously irradiated, that can be accurately measured at baseline.
* had no prior therapy with a selective MET inhibitor.
* no coinciding malignancy that would impact on survival.
* no metastasis limited to the bone only.

Module 2:

Patients recruited into Part A and Part B cohorts must have:

* tumours that are EGFR gene mutant that are currently progressing on treatment with a small molecule EGFR-TKI. Enrolment must be restricted to patients that are resistant to all relevant EGFR TKI therapy according to their tumour mutated status.
* received the EGFR-TKI as monotherapy for at least 12 weeks.
* tolerated their current dose of EGFR-TKI for at least 12 weeks.
* tumours that are MET gene amplified.
* had no prior therapy with a selective MET inhibitor.
* had no prior EGFR-TKI treatment of >2 lines.
* no past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* no significant GI disorders with diarrhoea as a major symptom e.g., Crohn's disease, mal-absorption, or CTCAE Grade >1 diarrhoea of any aetiology at the enrolment.
* no contra-indications (as per the relevant medication package insert) for therapy with the EGFR-TKI routinely used by their oncology unit.

In addition, patients recruited into Module 2 Part B cohorts must have:

* at least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with CT or MRI and which is suitable for accurate repeated assessment.
* no coinciding malignancy that would impact on survival.
* no metastasis limited to the bone only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events including dose-limiting toxicities | Baseline (C1D1) until 28 days after last administration of OMO-1
  The proportion of patients with treatment-emergent (serious) adverse events including dose-limiting toxicity (DLT)
Incidence of clinically significant abnormal measurements in physical examination, ophthalmological examination, vital signs, electrocardiogram (ECG), pregnancy test, lab tests and ECOG performance status | Screening until 28 days after last administration of OMO-1
  Physical examination and ophthalmological examination, vital signs; electrocardiogram (ECG); pregnancy test; haematology; clinical chemistry; urinalysis; plasma/renal makers; tumour markers; ECOG performance status

SECONDARY OUTCOMES:
Objective Response Rate | Screening until 28 days after last administration of OMO-1
  Objective response rate (ORR) by RECIST 1.1 - the proportion of patients with a confirmed reduction in tumour burden of a predefined amount (this will include short lived responses).
Percentage change in tumour size | Screening until 28 days after last administration of OMO-1
  Percentage change in tumour size will be determined for patients with measurable disease at baseline and is derived at each visit by the percentage change from baseline in the sum of the diameters of target lesions. The best percentage change in tumour size will be the patient's value representing the largest decrease (or smallest increase) from baseline in tumour size.
Maximal OMO-1 plasma concentration Cmax | Baseline (C1D1) and D1 in even cycles (C) until end of treatment (Part A) ; Baseline and C2D1 (Part B)
  Measurement of OMO-1 levels in plasma over time to calculate Cmax
Area under the OMO-1 plasma concentration curve (AUC) | Baseline (C1D1) and D1 in even cycles (C) until end of treatment (Part A) ; Baseline and C2D1 (Part B)
  Measurement of OMO-1 levels in plasma over time to calculate AUC
'Proof of mechanism' and 'proof of principle' pharmacodynamic biomarkers, including markers of tumour cell proliferation and apoptosis. | Screening until end of treatment
  Measurement of levels of 'Proof of mechanism' and 'proof of principle' pharmacodynamic biomarkers, including markers of tumour cell proliferation and apoptosis.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Lolkema, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (11):
- Mary Crowley Cancer Research, Dallas, Texas, United States
- University Hospital Antwerp, Edegem, Belgium
- France (3):
  - Institut Bergonie, Bordeaux
  - Hôpital La Timone, Marseille
  - lnstitut Gustave Roussy, Villejuif
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - UMCU Universitair Medisch Centrum Utrecht, Utrecht
- United Kingdom (4):
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - University of Oxford, Department of Oncology, Oxford

IPD SHARING:
Plan to Share IPD: No